CLINICAL TRIAL: NCT06423157
Title: Efficacy of a Plyometric and Stability Exercise Protocol in Female Basketball Players. A Controlled Clinical Study.
Brief Title: Plyometric and Stability Exercise Protocol in Female Basketball Players
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad Católica San Antonio de Murcia (Other)
Responsible Party: Principal Investigator, Rubén Cuesta-Barriuso, PhD, Principal Investigator, Universidad Católica San Antonio de Murcia
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: PlyoBask
Record Dates: First submitted 2024-05-15; First posted 2024-05-21 (Actual); Last update posted 2025-03-25 (Actual); Status verified 2024-05

CONDITIONS: Sports Physical Therapy
Keywords: Basketball; Plyometric Exercises; Stability; Flexibility; Agility; Physiotherapy
MeSH Terms: interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Three assessments will be made throughout the study: before the intervention (T0), after the experimental phase (T1) and after a 6-week follow-up period (T2). All variables will be assessed by an evaluator blinded to the assignment of the athletes to the study groups.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Experimental): The intervention period will last 6 weeks, with a periodicity of 2 weekly sessions of 20 minutes each. All interventions will take place at the Palacio de los Deportes de Murcia. All interventions will be carried out by the same physiotherapist, following the same protocol.
  The intervention of the experimental group will consist of a protocol using plyometric and stability exercises.
  Interventions: Other: Intervention
- Control group (No Intervention): The athletes included in the control group will not undergo any intervention and will continue with their usual routine.

INTERVENTIONS:
Other: Intervention — The intervention period will last 6 weeks, with a periodicity of 2 weekly sessions of 20 minutes each. All interventions will take place at the Palacio de los Deportes de Murcia. All interventions will be carried out by the same physiotherapist, following the same protocol. The intervention of the experimental group will consist of a protocol using plyometric and stability exercises.
  Arms: Experimental group

SUMMARY:
Introduction. Basketball is a high intensity intermittent sport, requiring jumping, running, accelerations and decelerations with changes of direction and lateral movements. Plyometric exercises are a training technique that consists of a cycle of muscle stretching and shortening in which the energy stored in the eccentric phase (lengthening) is released facilitating the production of maximum power in the concentric phase (shortening).

Objective. To analyse the efficacy of a physiotherapy intervention through a protocol of plyometric and stability exercises in the improvement of vertical jump, stability, flexibility and agility in federated female basketball players. The primary variable will be the vertical jump (My jump 2.0). Secondary variables will be stability (Y balance test), flexibility (Sit and Reach) and agility (T-Test).

Methods. Controlled, single-blind clinical study. 20 athletes will be randomised to the experimental and control groups. The intervention of the experimental group will consist of a protocol using plyometric and stability exercises. The athletes included in the control group will not perform any intervention and will continue with their usual routine. The intervention period will last 6 weeks, with a periodicity of 2 weekly sessions of 20 minutes each.

ELIGIBILITY:
Inclusion Criteria:

* Female players over 18 years of age.
* That during the study period they play basketball competing in the 1st Women's Division 1 category of the Basketball Federation of the Region of Murcia.
* That they perform strength exercises at least once a week.
* That they sign the informed consent document.

Exclusion Criteria:

* Players with knee or ankle injuries in the 6 months prior to the study.
* Players who use ankle or knee braces regularly.
* Players with lower limb surgery in the last year.
* Players whose participation is contraindicated by the team doctor, physiotherapist or physical trainer.

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2024-05-19 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Assess the changes in vertical jump | Screening visit, within the first seven days after treatment and after six weeks follow-up
  The vertical jump will be measured with the My jump 2.0® application. The athlete will be asked to jump as high as possible from a standing position, raising the body in the air by means of an impulse generated by the leg muscles. The evaluation consists of the recording of the jump, the calculation of the height of the vertical jump and the athlete's strength and speed levels. The unit of measurement of this tool is the centimetre, where the greater the distance, the higher the vertical jump.

SECONDARY OUTCOMES:
Assess the changes in stability | Screening visit, within the first seven days after treatment and after six weeks follow-up
  Stability is measured using the Y balance test. Three strips of adhesive tape are placed on the floor in a Y shape. The athlete, placed in the centre of the Y, will maintain unipodal balance while with the contralateral leg trying to reach the farthest point in each direction (anterior, posteromedial and posterolateral), without lifting the heel of the supporting foot which is the one being evaluated. Three attempts shall be made with each leg. The distance is measured with a tape measure, in centimetres (19), where the greater the distance, the greater the stability.
Assess the changes in flexibility | Screening visit, within the first seven days after treatment and after six weeks follow-up
  Flexibility will be assessed with the Sit and Reach test. The athlete will sit on the floor, with her knees straight and her feet placed against the edge of a box. From this position, the participant shall progressively perform a trunk flexion, trying to reach as far as possible with the tips of her hands on the scale graduated in centimetres on the box. The unit of measurement for this test is the centimetre, where the greater the distance reached, the greater the flexibility.
Assess the changes in agility | Screening visit, within the first seven days after treatment and after six weeks follow-up
  Agility will be assessed with the T-Test. Four cones should be placed in a T-shape: A at the starting point; B at 9.14 m forward; and C and D at the sides of this at 4.57 m the other two cones. The athlete must go as fast as possible to cone B and touch it with the tip with her right hand, then she must go to the sides touching cones C and D with the hand of the same side, return to touch cone B with the left hand and lastly, move backwards and go over cone A. The unit of measurement is the second, where lower times indicate efficient agility.

CONTACTS AND LOCATIONS:
Locations (1):
- Universidad Católica San Antonio, Murcia, Murcia, Spain